CLINICAL TRIAL: NCT02271139
Title: An Open Label, Multicenter, Single-Arm, Expanded Access Study of Alectinib for Patients With ALK-Rearranged Non-Small Cell Lung Cancer After Disease Progression on or Intolerance to Prior ALK Tyrosine Kinase Inhibitor Therapy
Brief Title: Expanded Access Study of Alectinib for Participants With Anaplastic Lymphoma Kinase (ALK)-Rearranged Non-Small Cell Lung Cancer (NSCLC) After Disease Progression on or Intolerance to Prior ALK Tyrosine Kinase Inhibitor Therapy
Status: No longer available | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29453
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

INTERVENTIONS:
Drug: Alectinib — Alectinib 600 mg administered orally with food.

SUMMARY:
This is an open-label, multicenter, single-arm, expanded access study designed to provide alectinib to participants with ALK-rearranged NSCLC after disease progression on or intolerance to prior ALK tyrosine kinase inhibitor (TKI) therapy. Participants will receive alectinib until disease progression, unacceptable toxicity, withdrawal of consent, patient or physician decision to discontinue treatment, death, alectinib becomes commercially available in the United States following approval of alectinib by the FDA, or the Sponsor decides to close the trial, whichever occurs first (approximately 15 months).

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced (American Joint Committee on Cancer [AJCC] Stage IIIB) not amenable to curative therapy or metastatic (AJCC Stage IV) NSCLC
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-3
* Histologically confirmed NSCLC
* Documented ALK rearrangement as assessed by approved fluorescence in situ hybridization (FISH) test, using the Vysis ALK Break Apart FISH Probe Kit or the Ventana immunohistochemistry (IHC) test
* After disease progression on or intolerance to prior ALK TKI therapy: 1) participants need to have a minimum washout period of at least 5 half-lives between the last dose of ALK TKI therapy or other targeted therapies and the first dose of study treatment; 2) participants must have recovered from treatment toxicities to less than or equal to (</=) Grade 1 or to their pretreatment levels (for participants who have developed interstitial lung disease [ILD], they must have fully recovered); 3) participants can either be chemotherapy-naïve or have received at least one line of platinum-based chemotherapy for locally advanced or metastatic disease
* Recovery from effects of any major surgery or significant traumatic injury at least 28 days before the first dose of study treatment
* Adequate hematological and renal function
* Agreement to use highly effective methods of contraception per protocol definitions

Exclusion Criteria:

* Prior therapy with alectinib
* Participants with symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of steroids within 1 week prior to Day 1 to manage CNS symptoms
* Administration of strong/potent cytochrome P450 3A (CYP3A) inhibitors or inducers, or agents with potential QT prolonging effects within 14 days prior to first administration of study drug
* Participants with liver disease
* Any clinically significant concomitant disease or condition that could interfere with the conduct of the study
* Active or uncontrolled infectious diseases requiring treatment
* History of organ transplant
* Participants with baseline QTc > 470 milliseconds (ms) or participants with symptomatic bradycardia
* Pregnant or lactating, or intending to become pregnant during the study
* History of hypersensitivity to any of the additives in alectinib formulation
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the participants before trial entry
* Serious, uncontrolled infections or current known infection with human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (45):
  - University of Alabama, Bimingham, Alabama
  - Southern Cancer Center, Daphne, Alabama
  - Southern Cancer Center, Mobile, Alabama
  - Southern Cancer Center - Mobile, Mobile, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Lalita Pandit Inc., Fountain Valley, California
  - University of California San Diego Medical Center; Moores Cancer Center, La Jolla, California
  - Loma Linda Cancer Center, Loma Linda, California
  - LAC USC Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - St. Joseph Heritage Healthcare, Sebastopol, California
  - Innovative Clinical Research Institute, Whittier, California
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - Loyola University Med Center, Maywood, Illinois
  - Investigative Clin Rsch of IN, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Partners Can Ctr, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr; Hem/Onc, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute - Farmington Hills/Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Comprehensive Cancer Care, P.C., St Louis, Missouri
  - Billings Clinic Cancer Center; Billings Cancer Research, Billings, Montana
  - San Juan Oncology Associates, Farmington, New Mexico
  - Columbia University Medical Center; Clinical Research Management Office, New York, New York
  - W.G. Bill Hefner VA Medical Center, Salisbury, North Carolina
  - Mark H. Zangmeister Center, Columbus, Ohio
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Oregon Health & Science Uni, Portland, Oregon
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Cancer Treatment Centers of America - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - West Penn Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina; Hollings Cancer Center, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin; Oncology, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sikkema BJ, Baart SJ, Paats MS, Smit EF, Schols AMWJ, Mathijssen RHJ, van Rossum EFC, Dingemans AC. Body Weight Gain Associated With Alectinib in Patients With ALK+ Non-Small Cell Lung Cancer: Pooled Analysis of Individual Patient Data From Four Prospective Clinical Trials. J Clin Oncol. 2025 Feb 20;43(6):641-650. doi: 10.1200/JCO-24-01579. Epub 2024 Dec 11. PMID 39661917